CLINICAL TRIAL: NCT04844788
Title: A Consensus on Opioid Prescription for Oncologic Patients in Latin America - A DELPHI Study.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Felipe Porto Rangel, Dr, Hospital Sirio-Libanes
Other Study IDs: 08042021
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Cancer Patients; Cancer-related Pain
Keywords: opioids; cancer-related pain; end-of-life; opioid abuse
MeSH Terms: conditions — Cancer Pain; Death; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As seen worldwide, cancer incidence is increasing in Latin America achieving an amount of 1.3 million new cases annually.1 In addition, it is expected that up to 70% of patients with cancer will experience pain2, one of the most distressing symptoms in patients with advanced cancer.

And despite of advances in cancer therapies, opioids remain the mainstay treatment of cancer-related moderate-to-severe and end-of-life pain.3 However, concerns regarding opioid prescriptions have emerged for reasons like the risk of misuse and the possibility of cancer progression.

In the last decades, an increase in consumption of opioids as well as in opioids-related deaths generating the so called 'opioid crisis'. This rise is mainly due to abuse / addiction of opioids. Consequently, oncologic patients are at risk for abuse, as well as for aberrant use, which can complicate the course of cancer treatment.4 5 Another feature of opioids use in cancer patients is that it may contribute to disease progression. Experimental studies suggest that opioids can may lead to immunosuppression and tumor progression or recurrence.6-8 On the other hand, retrospective analysis of clinical data shows conflicting results and trials are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Head of anesthesia, Pain management and palliative care departments of cancer hospitals in Latin America.

Exclusion Criteria:

* Surveys not answered.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The experts assessed in this study will be the heads of anesthesia, pain management and palliative care of leading cancer hospitals of Latin America countries. For each Latin America country will be assessed 3 experts maximum.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Survey answers | Up to 3 (three) months
  answers of the survey sent

CONTACTS AND LOCATIONS:
Overall Officials: Felipe P Rangel, PhD, Principal Investigator — MD Anderson; Juan P Cata, PhD, Study Director — M.D. Anderson Cancer Center
Locations (1):
- Felipe Porto Rangel, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared. The data collected will be summarized and a consensus of the answers of all participants will reported.